CLINICAL TRIAL: NCT04319432
Title: Optimal Duration of Voice Rest Voice Following Phonosurgery for Benign Vocal Lesions: Prospective Randomized Study.
Brief Title: Optimal Duration of Voice Rest After Surgery for Benign Vocal Lesions
Acronym: VR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TASMC20YOK037218CTIL
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Vocal Fold Polyp; Vocal Cord Cyst; Vocal Nodules in Adults

STUDY DESIGN:
Intervention Model Description: Prospective Study. In this study, patients will be placed into one of two different groups of voice rest duration. The voice rest durations will last either 3 or 7 days. Voice recording results of the different groups will be examined and analyzed. At the conclusion of this study, we hope to provide some clarity as to the optimal duration of voice rest following phonosurgery.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 days voice rest (Experimental)
  Interventions: Behavioral: Voice rest
- 7 days voice rest (Experimental)
  Interventions: Behavioral: Voice rest

INTERVENTIONS:
Behavioral: Voice rest — The first days will take place in hospitalization to assess patient complience to voice rest. Patients will be instructed to continue voice rest at home up to 7 days accourding to group allocation in the study. The confirmation of voice rest will relay on patient report (telephonic approval), after the voice rest period will end.

SUMMARY:
Aim of Study:

To determine the optimal duration of voice rest following phonosurgery for patients who undergo phonosurgery due to benign vocal cord lesions IE: vocal fold nodules, cysts, polyps, granulomas, leukoplakia, and subepithelial edema.

DETAILED DESCRIPTION:
Optimal Duration of Voice Rest Voice Following Phonosurgery for benign vocal lesions: Prospective Randomized Study

Background:

Phonosurgery is performed in order to improve voice quality in patients with various vocal fold pathologies including nodules, cysts, polyps, granulomas, leukoplakia, and subepithelial edema. It is customary to order the patients voice rest following vocal fold surgery, however, according to the current literature, it is not well known how long patients should remain in voice rest following phonosurgery (regardless of the type of benign lesion) in order to achieve the best voice quality results. In the literature, there is one preliminary study that shows that when voice quality was assessed at 15 days post-surgery, patients with voice rest of 10 days had better voice outcomes compared to patients with 5 days voice rest(1). A contradicting study, that measured voice outcomes in patients at 1, 3, and 6 months post-operatively, shows that a short voice rest of 3 days lead to better voice results compared to a 7 days voice rest(2).

The aim of our study is to determine the optimal duration (3 versus 7 days) of voice rest following phonosurgery for patients who undergo phonosurgery due to benign vocal cord lesions in order to achieve better voice quality post-operatively. In this study, patients will be randomly assigned into one of 2 different groups of voice rest durations: either 3 or 7 days following surgery. Patients will undergo pre and post (at 1, 3 and 6 months) operative voice testing. Voice quality testing will include: perceptual voice analysis using the GRABS (grade, roughness, asthenia, breathiness, and strain) scale, Voice Handicap Index-10 (VHI) questionnaire, measurement of maximum phonation time (MPT), and computerized voice analysis including voice intensity, fundamental frequency (F0), jitter, shimmer, and dysphonia severity index (DSI).

ELIGIBILITY:
Inclusion Criteria:

* • Patients who undergo phonosurgery for benign vocal fold lesions.

  * Adults (18-90years).
  * Patients who can provide and give informed consent.

Exclusion Criteria:

* • Patients without a complete medical record

  * Patients who are unable or unwilling to give informed consent
  * Patients younger than 18 years of age or older then 90 years
  * Patients who are pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-12 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
better voice quality by GRABS scale | 6 months post op
  GRABS scale- Grade, Roughness, Breathiness, Asthenia, Strain (GRBAS) each ranked from 0 to 3

CONTACTS AND LOCATIONS:
Overall Officials: Yael Oestreicher kedem, MD, Principal Investigator — TASMC
Locations (1):
- TASMC, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
Anonymization of study patients Patient information (I.e. name, ID number, etc.) will be collected and kept confidential throughout the study so that the patients cannot be re-traced or identified. The information will be gathered by the main investigator kept in an encrypted file with a password required for access on the main researcher's computer. Information will not be sent or distributed outside the hospital to anyone.